CLINICAL TRIAL: NCT05456386
Title: BioRhythm Health Coaching and Sleep Monitoring Program for Weight Loss
Brief Title: The BioRythm Guided Weight Loss Study Will Test a Novel Behavioral Health Intervention Combined With Fitbit Technology Monitoring in Obese Individuals to Determine if it Promotes Weight Loss, Improves Objective Measures of Sleep Health, and Aids in Developing a Consistent Mealtime Routine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stephen Hutchison (Other)
Responsible Party: Sponsor-Investigator, Stephen Hutchison, Research Coordinator, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIORHYTHMSTUDYTBD
Record Dates: First submitted 2022-07-06; First posted 2022-07-13 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Circadian Rhythm Approach to Weight Loss (CRAWL) Intervention Arm (Experimental): The Circadian Rhythm Approach to Weight Loss (CRAWL) intervention subjects will continuously wear their Fitbit Versa 2 (aside from periodic charging periods) and participate in the pre-scheduled CRAWL sessions. Every week, subjects will complete a sleep diary, which assesses subject's time in bed, sleep latency, awakenings, wake after sleep onset, awakening time, overall sleep quality, overall refreshed rating, naps, exercise, energy level and mood. Subjects are to ensure their Fitbit is sufficiently charged every night before bed and they are to wear their Fitbit continuously throughout the night. Subjects will weigh themselves using their home scale each week prior to exercise, taking a shower or eating breakfast. They will record their weight in their provided weight tracking sheet
  Interventions: Behavioral: The Circadian Rhythm Approach to Weight Loss (CRAWL)
- Waitlist Control Arm (No Intervention): Waitlist control subjects will follow the same protocol outlined above for 16 weeks minus the scheduled CRAWL sessions. When the initial treatment arm has completed their 16 weeks of group sessions, the waitlist control group will begin their CRAWL sessions.

INTERVENTIONS:
Behavioral: The Circadian Rhythm Approach to Weight Loss (CRAWL) — The Circadian Rhythm Approach to Weight Loss (CRAWL) is a behavioral intervention that is designed to provide support for behavioral change to improve sleep and feeding parameters that will lead to sustainable weight loss.
  Arms: The Circadian Rhythm Approach to Weight Loss (CRAWL) Intervention Arm

SUMMARY:
The BioRhythm study will test a novel behavioral health intervention that utilizes personalized behavioral health counseling as well as sleep and activity data obtained via wearable technology to promote weight loss in obese individuals.

1. Determine whether the use of the The Circadian Rhythm Approach to Weight Loss (CRAWL) intervention results in improvements in weight loss and a reduction in mean daily eating opportunity window.

   a. Hypothesis: Compared to a wait list control, the CRAWL intervention will induce greater changes in weight loss and body mass index and mean daily eating opportunity window.
2. Establish whether use of the CRAWL intervention results in changes in objectively estimated circadian rhythm, activity levels, sleep duration, sleep architecture, and sleep timing.

   1. Hypothesis: Compared to a wait list control, the CRAWL intervention will induce improvements in all metrics described above.

DETAILED DESCRIPTION:
Subjects interested in the participation of this study will be directed to a screening questionnaire to determine study eligibility. Eligible participants will be contacted by the study coordinator to schedule a virtual meeting to complete the informed consent procedure.

Upon the completion of the informed consent procedure, subjects will be mailed a Fitbit Versa 2 and instructions for use. Subjects will be asked to contact the study team when they receive their devices to schedule a virtual teleconference to walk them through detailed use instructions as well as data uploading procedures on their mobile device. The study team will be able to address any concerns or questions at this time. Subjects will also be reminded that they may contact the study team at any time if they have questions or concerns.

The Fitbit Vera 2 is a wristband that includes sensors for heart rate and accelerometry. From these sensors, data such as resting heart rate, activity patterns, and sleep continuity and architecture can be extracted. These wristbands are worn continuously and charged every 7 days. Data are synced to an app that the subject will install on their mobile device. The app will give health tips for the patient to improve sleep, activity, and nutrition and then send monitoring information to the study team.

Prior to using the device, the subject will have a pre-scheduled consultation with a designated health aide via virtual conference to introduce the weight loss program. The health aide will also complete a structured interview during this consultation which will include a series of questionnaires.

After subjects have been oriented to the devices and have completed their preliminary intake questionnaires and medical history, they will begin the following protocol:

Subjects will be randomly assigned to a waitlist control group or the The Circadian Rhythm Approach to Weight Loss (CRAWL) intervention group. The wait list control group serves as a benchmark, allowing for the comparison of the CRAWL intervention to a control group to evaluate the intervention's impact. This will allow for the assessment of the intervention's efficacy against not receiving treatment during that same time period (while still providing all participants with treatment eventually).

Subjects assigned to the treatment arm will be scheduled for a total of 10 CRAWL group sessions over 16 weeks with a designed study member that will last approximately 1 hour.

A CRAWL health coach will assess each subject's individual chronotype (via the Munich Chronotype Questionnaire) to develop a preliminary time-restricted feeding (TRF) regimen. For example, a subject that scores as a "morning" type will be counseled to adhere to an eating window that starts earlier in the day (e.g., 8am to 4pm). This regimen will be further refined based on the subjective feedback of the subject as well as objective Fitbit data. Eating windows will also be developed around cases in which subjects are prescribed medications that are commonly taken with meals (e.g., metformin).

The connection between nutrition and circadian rhythm will be addressed in the CRAWL sessions, however, subjects will not be specifically encouraged to adhere to any one macronutrient schema. Instead, discussions will revolve around the resolution of potential problematic eating patterns as well as the avoidance of processed, packaged foods. Nutritional supplements will be permitted throughout the course of the study as long as they are consumed within the defined feeding windows.

CRAWL intervention subjects will continuously wear their Fitbit Versa 2 (aside from periodic charging periods) and participate in the pre-scheduled CRAWL sessions. Every week, subjects will complete a sleep diary, which assesses subject's time in bed, sleep latency, awakenings, wake after sleep onset, awakening time, overall sleep quality, overall refreshed rating, naps, exercise, energy level and mood. Subjects are to ensure their Fitbit is sufficiently charged every night before bed and they are to wear their Fitbit continuously throughout the night. Subjects will weigh themselves using their home scale each week prior to exercise, taking a shower or eating breakfast. Subjects should then make sure that their Fitbit devices are synced correctly, and all data has been successfully uploaded to the study team. Subjects will be informed to contact the study team at any time if they encounter any technical problems with their devices.

Waitlist control subjects will follow the same protocol outlined above for 16 weeks minus the scheduled CRAWL sessions. When the initial treatment arm has completed their 16 weeks of group sessions, the waitlist control group will begin their CRAWL sessions.

Subject participation will last 16 weeks (32 weeks for the waitlist control subjects). After completion of the CRAWL intervention, subjects will then engage in a final virtual conference or in person meeting with the study team, in order to discuss their experiences with the study and to again complete a series of questionnaires provided at the start of the study. After completing this call and all study procedures, involvement in the study will be complete.

The BioRythm Guided Weight Loss project is a proof-of-concept pilot study designed to evaluate the potential efficacy of the CRAWL intervention to induce weight loss. The CRAWL intervention utilizes a multifactorial approach to achieve this goal. This pilot project does not have the budget nor the scope to determine whether and to what degree each aspect of the intervention induced weight loss (i.e., is time restricted feeding or improved sleep quality driving weight loss?). Future studies will be designed to dismantle the CRAWL intervention to determine the relative efficacy of each piece of the whole package.

Data will be collected and managed through the HIPAA compliant platform RevUP, supported by MD Revolution. As noted, due to the small sample size and limited scope, this study will likely be underpowered for statistical significance and will therefore focus primarily on descriptive rather than inferential statistics. Independent t-tests will be used to determine if there is a significant difference in primary and secondary outcomes between the CRAWL intervention and waitlist control groups. Paired t-tests will be performed to compare within-group differences of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 - 75 years old
2. Able to read and write fluently in English or Spanish
3. Access to a mobile device for video calls, online questionnaires, syncing devices, and communication with study staff
4. Access to a residential mailing address for shipping study materials
5. Body Mass Index (BMI) ≥ 30
6. Self-report that they have a problem with their weight that they wish to improve
7. Must be able to participate in mild to moderate physical activity
8. Access to a mechanical or digital scale

Exclusion Criteria:

1. Have a severe, untreated sleep disorder (e.g., Obstructive Sleep Apnea (OSA), Restless Leg Syndrome (RLS), insomnia, narcolepsy)
2. Patients who are unable to participate in prolonged fasting periods such as insulin dependent diabetics.
3. Have a medical condition that would interfere with their ability to complete all study procedures or would render measurements invalid (e.g., some autoimmune conditions, cardiac conditions, endocrine conditions, or chronic pain conditions)
4. Unable to achieve a regular sleep schedule, where bed and wake times are kept within a 2-hour window 7 days per week
5. Unable to maintain a regular sleep schedule during the night, beginning no earlier than 9pm and ending no later than 10am
6. Have not engaged in shift work for the past month, and will refrain from shift work during the study
7. Are unable to restrict alcohol consumption to no more than 2 drinks within 4 hours of sleep
8. Are unable to restrict caffeine use to no coffee or caffeinated beverages after 12pm during the study
9. Regularly smoke or use other tobacco products
10. Are unable to restrict cannabis products (e.g., marijuana) or cannabis-derived medicinal products (e.g., Marinol) within 4 hours of sleep
11. Are pregnant
12. Are a full-time caregiver to an individual that requires attending during the evening and night
13. Physically disabled or confined to a bed, wheelchair, or walker.
14. Presence of a diagnosed eating disorder
15. Currently use prescription or over-the-counter appetite suppressants or other prescription drugs that may interfere with appetite (e.g., Adderall)
16. Are diagnosed with bipolar disorder, schizophrenia, or untreated depression (PHQ-9 > 15).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The Circadian Rhythm Approach to Weight Loss (CRAWL) Intervention Weight Loss | 4 months
  Change in recorded participant weight (kg).
The Circadian Rhythm Approach to Weight Loss (CRAWL) Intervention Daily Eating Opportunity Window | 4 months
  Change in mean daily eating opportunity window defined by the elapsed time between the consumption of the first meal of the day and the last meal of the day.

SECONDARY OUTCOMES:
The Circadian Rhythm Approach to Weight Loss (CRAWL) Intervention Total Sleep Time | 4 months
  Change in Fitbit estimated Total Sleep Time defined as the total amount of sleep time scored during the total recording time throughout the night.
The Circadian Rhythm Approach to Weight Loss (CRAWL) Intervention Sleep Architecture | 4 months
  Change in Fitbit estimated sleep stages defined as the total recorded amount of time spent in wake, N1, N2, N3, and rapid eye movement (REM) sleep throughout the night.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284
- [Background] Kahn SE, Hull RL, Utzschneider KM. Mechanisms linking obesity to insulin resistance and type 2 diabetes. Nature. 2006 Dec 14;444(7121):840-6. doi: 10.1038/nature05482. PMID 17167471
- [Background] Luppino FS, de Wit LM, Bouvy PF, Stijnen T, Cuijpers P, Penninx BW, Zitman FG. Overweight, obesity, and depression: a systematic review and meta-analysis of longitudinal studies. Arch Gen Psychiatry. 2010 Mar;67(3):220-9. doi: 10.1001/archgenpsychiatry.2010.2. PMID 20194822
- [Background] Clark I, Stucky B, Azza Y, Schwab P, Muller S, Weibel D, Button D, Karlen W, Seifritz E, Kleim B, Landolt HP. Diurnal variations in multi-sensor wearable-derived sleep characteristics in morning- and evening-type shift workers under naturalistic conditions. Chronobiol Int. 2021 Dec;38(12):1702-1713. doi: 10.1080/07420528.2021.1941074. Epub 2021 Jul 18. PMID 34278901
- [Background] Lujan MR, Perez-Pozuelo I, Grandner MA. Past, Present, and Future of Multisensory Wearable Technology to Monitor Sleep and Circadian Rhythms. Front Digit Health. 2021 Aug 16;3:721919. doi: 10.3389/fdgth.2021.721919. eCollection 2021. PMID 34713186
- [Background] Kolla BP, Mansukhani S, Mansukhani MP. Consumer sleep tracking devices: a review of mechanisms, validity and utility. Expert Rev Med Devices. 2016 May;13(5):497-506. doi: 10.1586/17434440.2016.1171708. Epub 2016 Apr 18. PMID 27043070
- [Background] Majumder S, Mondal T, Deen MJ. Wearable Sensors for Remote Health Monitoring. Sensors (Basel). 2017 Jan 12;17(1):130. doi: 10.3390/s17010130. PMID 28085085
- [Background] Ong JL, Lau T, Massar SAA, Chong ZT, Ng BKL, Koek D, Zhao W, Yeo BTT, Cheong K, Chee MWL. COVID-19-related mobility reduction: heterogenous effects on sleep and physical activity rhythms. Sleep. 2021 Feb 12;44(2):zsaa179. doi: 10.1093/sleep/zsaa179. PMID 32918076
- [Background] Chinoy ED, Cuellar JA, Huwa KE, Jameson JT, Watson CH, Bessman SC, Hirsch DA, Cooper AD, Drummond SPA, Markwald RR. Performance of seven consumer sleep-tracking devices compared with polysomnography. Sleep. 2021 May 14;44(5):zsaa291. doi: 10.1093/sleep/zsaa291. PMID 33378539
- [Background] Roberts LM, Jaeger BC, Baptista LC, Harper SA, Gardner AK, Jackson EA, Pekmezi D, Sandesara B, Manini TM, Anton SD, Buford TW. Wearable Technology To Reduce Sedentary Behavior And CVD Risk In Older Adults: A Pilot Randomized Clinical Trial. Clin Interv Aging. 2019 Oct 23;14:1817-1828. doi: 10.2147/CIA.S222655. eCollection 2019. PMID 31695350
- [Background] Batsis JA, Petersen CL, Clark MM, Cook SB, Lopez-Jimenez F, Al-Nimr RI, Pidgeon D, Kotz D, Mackenzie TA, Bartels SJ. A Weight Loss Intervention Augmented by a Wearable Device in Rural Older Adults With Obesity: A Feasibility Study. J Gerontol A Biol Sci Med Sci. 2021 Jan 1;76(1):95-100. doi: 10.1093/gerona/glaa115. PMID 32384144
- [Background] Shechter A, Grandner MA, St-Onge MP. The Role of Sleep in the Control of Food Intake. Am J Lifestyle Med. 2014 Nov 1;8(6):371-374. doi: 10.1177/1559827614545315. Epub 2014 Aug 6. PMID 27065757
- [Background] Tahara Y, Shibata S. Chronobiology and nutrition. Neuroscience. 2013 Dec 3;253:78-88. doi: 10.1016/j.neuroscience.2013.08.049. Epub 2013 Sep 3. PMID 24007937
- [Background] Rynders CA, Thomas EA, Zaman A, Pan Z, Catenacci VA, Melanson EL. Effectiveness of Intermittent Fasting and Time-Restricted Feeding Compared to Continuous Energy Restriction for Weight Loss. Nutrients. 2019 Oct 14;11(10):2442. doi: 10.3390/nu11102442. PMID 31614992
- [Background] Chaix A, Lin T, Le HD, Chang MW, Panda S. Time-Restricted Feeding Prevents Obesity and Metabolic Syndrome in Mice Lacking a Circadian Clock. Cell Metab. 2019 Feb 5;29(2):303-319.e4. doi: 10.1016/j.cmet.2018.08.004. Epub 2018 Aug 30. PMID 30174302
- [Background] Arble DM, Bass J, Laposky AD, Vitaterna MH, Turek FW. Circadian timing of food intake contributes to weight gain. Obesity (Silver Spring). 2009 Nov;17(11):2100-2. doi: 10.1038/oby.2009.264. Epub 2009 Sep 3. PMID 19730426
- [Background] Galindo Munoz JS, Gomez Gallego M, Diaz Soler I, Barbera Ortega MC, Martinez Caceres CM, Hernandez Morante JJ. Effect of a chronotype-adjusted diet on weight loss effectiveness: A randomized clinical trial. Clin Nutr. 2020 Apr;39(4):1041-1048. doi: 10.1016/j.clnu.2019.05.012. Epub 2019 May 21. PMID 31153674